CLINICAL TRIAL: NCT00589212
Title: A Phase II Study Utilizing Focal Radiation in Patients With 1-3 Brain Metastases
Brief Title: GliaSite 1-3 Mets Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Collaborators: Methodist Healthcare (Other)
Responsible Party: Allen K. Sills, Jr. MD, University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-700; NCT00096252 (obsolete NCT alias)
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Brain Metastases
Keywords: GliaSite; Brain metastases; 1-3 METS
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients with 1-3 brain metastases
  Interventions: Device: GliaSite Radiation Therapy System

INTERVENTIONS:
Device: GliaSite Radiation Therapy System — GliaSite RTS is designed to deliver intracavitary radiation therapy for brain tumors. Following surgical resection, the balloon catheter is inflated to fill the cavity and Iotrex radiotherapy solution infused. It is a single applicator system that provides a uniform and conformal dose to the resection cavity.

SUMMARY:
This study has been designed to compile information on the efficacy of the GliaSite RTS combined with radiosurgery in the treatment of newly diagnosed metastatic brain tumors.

DETAILED DESCRIPTION:
Data relevant to the evaluation the effectiveness of the GliaSite RTS for a resected dominant brain metastases will be collected. The GliaSite RTS is a radionuclide applicator and liquid radionuclide (Iotrex) designed to deliver intracavitary radiation therapy for resected brain tumors. In this case, it will irradiate the resected margins. Brain metastases not surgically removed will be then treated with radiosurgery

ELIGIBILITY:
Inclusion Criteria:

* Have 1-3 newly diagnosed supratentorial metastatic brain lesions with at least one being dominant and eligible for surgical resection as visualized on enhanced MRI scan
* Have histological evidence of metastatic carcinoma on intraoperative pathology (frozen section) or final pathology report
* Have a Karnofsky Performance Status (KPS) >=70
* Have systemic disease which is judged to be stable and has been staged within the last 6 weeks
* Have a life expectancy of >= 6 month, based upon extent of systemic disease
* Be at least 18 years of age Give informed consent (or have legal representative give informed consent)

Exclusion Criteria:

* Be receiving or have plans to receive conventional or investigational systemic agents for the metastatic brain tumor.
* Be receiving or have plans to receive external beam radiation therapy to the brain.
* Have received prior conventional or investigational systemic agents, including the use of Gliadel Wafers or Temodar, for the treatment of the brain metastasis.
* Be pregnant or breast-feeding.
* Have uncontrolled hypertension, unstable angina pectoris, evidence of uncontrolled cardiac dysrhythmia.
* Have other serious concurrent infection or other medical illness which would jeopardize the ability of the patient to safely undergo resection and brachytherapy.
* Have histology of lymphoma or small-cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is to evaluate the 6 month and 1 year local control rate for 1-3 brain metastases treated with intracavitary radiation therapy. | Data collected at the time of implant, within 72 hours of implant, pre-brachytherapy, brachytherapy, radiosurgery, 1 and 3 months post brachytherapy and every 3 months thereafter

SECONDARY OUTCOMES:
Overall survival, distant brain recurrence, toxicity and quality of life. | Survival

CONTACTS AND LOCATIONS:
Overall Officials: Allen K Sills, Jr., MD, Principal Investigator — University Hospital
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States